CLINICAL TRIAL: NCT03340233
Title: A New Framework for Understanding the Mechanism of Diastolic Dysfunction
Brief Title: Understanding the Mechanisms of Diastolic Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI left the institution and closed the study prior to enrolling any participants
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Ennis, PhD, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#17-000695; 1R01HL131823-01A1 (NIH)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Healthy
Keywords: diastolic dysfunction; mechanism; MRI magnetic resonance imaging; ejection fraction
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Group 1 includes 25 healthy subjects recruited in Year 1 to undergo cardiac MRI without contrast.
  Interventions: Diagnostic Test: MRI (cardiac)
- Group 2 (Experimental): Group 2 includes 25 healthy subjects recruited in Year 2 to undergo cardiac MRI without contrast.
  Interventions: Diagnostic Test: MRI (cardiac)
- Group 3 (Experimental): Group 3 includes 33 patients with Heart Failure with Preserved Ejection Fraction (HFpEF) who will undergo cardiac MRI at baseline and at six months to assess diagnostic sensitivity of MRI measurement.
  Interventions: Diagnostic Test: MRI (cardiac) off-label use gadolinium contrast (IND exempt)

INTERVENTIONS:
Diagnostic Test: MRI (cardiac) off-label use gadolinium contrast (IND exempt) — Clinical MRI
  Arms: Group 3
Diagnostic Test: MRI (cardiac) — MRI without contrast
  Arms: Group 1; Group 2

SUMMARY:
Heart failure is a clinical syndrome marked by breathlessness, even at low levels of exertion, general fatigue, and fluid retention and is estimated to affect 5.1 million people in the United States. Heart failure with preserved ejection fraction (HFpEF) means that the heart pumps enough blood to the body, but patients still have terrible symptoms. It is estimated to account for about 50% of all heart failure cases. Experts agree that impaired filling of the heart, perhaps due to "stiffness" of the heart muscle itself, critically underlies HFpEF. There is currently no clinical technique for measuring heart muscle (myocardial) stiffness; the very definition of "myocardial stiffness" remains poorly established. Consequently, the ability to study the mechanisms that underlie HFpEF is virtually non-existent, and limited treatment options will persist without significant advances. The objective of this project is to use an Equilibrium-Material-Stability (EMS) framework that couples patient-specific clinical MRI and heart pressure data in a computational model of the heart to diagnose changes in myocardial stiffness. The central hypothesis is that the new EMS framework for understanding the mechanisms of diastolic dysfunction in HFpEF will be more sensitive and outperform currently available approaches.

DETAILED DESCRIPTION:
The study has three aims. The first aim of the project is to refine MRI techniques using "free-breathing" versus "breath-holding" measurements. Twenty-five normal volunteers will undergo MRI to refine "free-breathing" cardiac imaging and enable construction of patient-specific computer models of the heart. The second aim of the project is to validate and test the myocardial stiffness evaluation framework derived through the first objective in human subjects. Twenty-five normal volunteers will undergo MRI and the data from these images will be compared to specially constructed 3D printed models of the heart, enabling refinement of the EMS framework to separate structural stiffness from material stiffness. The third aim of the project is to measure changes in myocardial stiffness in patients with HFpEF. Thirty-three subjects with current diagnostic criteria for HFpEF will be evaluated at baseline and at six months to evaluate myocardial stiffness and cardiac MRI biomarkers. Specifically, this aim will establish the diagnostic sensitivity of the EMS framework with comparison to cardiac MRI biomarkers of increased stiffness, thereby providing mechanistic insight to one critical underlying cause of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

1. Healthy adults

Patients with Heart Failure with Preserved Ejection Fraction

1. Patient scheduled for catheterization at UCLA Medical Center
2. Ejection fraction >/= 50%
3. Signs and symptoms of heart failure
4. Excluded other potential non-cardiac etiologies of heart failure

Exclusion Criteria:

Healthy volunteers

1. Known medical condition that impacts heart health
2. Contraindications to MRI (e.g., pacemaker/ICD, or claustrophobia)

Patients with Heart Failure with Preserved Ejection Fraction

Exclusion Criteria:

1. Contraindications to MRI (e.g., pacemaker/ICD, or claustrophobia)
2. Prior MI or history of PCI/CABG
3. Worse than mild valvular disease
4. Any indication for ICD implantation
5. Contraindication to MRI contrast agents or eGRF <30 ml/min/1.73m2 or MRI exams (e.g., pacemaker/ICD or claustrophobia).
6. Atrial fibrillation or unstable cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of the EMS framework with comparison to cardiac MRI biomarkers of increased stiffness, thereby providing mechanistic insight to one critical underlying cause of HFpEF. | Five years
  Assess the diagnostic sensitivity of MRI method by analyzing baseline and six month longitudinal characteristics in myocardial stiffness measured in patients with HFpEF

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Ennis, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No